CLINICAL TRIAL: NCT06151782
Title: Towards Comprehensive Analytical Methods for Partially Hydrolysed Gluten to Assess Product Safety for Celiac Disease Patients
Brief Title: Immunosafe-CeD: Are Partially Hydrolysed Gluten Harmful to Celiac Disease Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Knut E. A. Lundin, Senior consultant, professor, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2637128
Record Dates: First submitted 2023-11-14; First posted 2023-11-30 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Celiac Disease; Food Intolerance
MeSH Terms: conditions — Celiac Disease; Food Intolerance | interventions — Glutens

STUDY DESIGN:
Intervention Model Description: Participants will be challenged by single bolus five times four weeks apart.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Wheat gluten (Active Comparator): In slurry, measurement of immune activation (Interleukin-2) four hours after intake
  Interventions: Dietary Supplement: Wheat gluten 1000 mg
- Barley gluten (Experimental): In slurry, measurement of immune activation (Interleukin-2) four hours after intake
  Interventions: Dietary Supplement: Barley gluten 1000 mg
- Low dose barley gluten (Experimental): In slurry, measurement of immune activation (Interleukin-2) four hours after intake
  Interventions: Dietary Supplement: Barley gluten 50 mg
- Low dose hydrolyzed barley gluten (Experimental): In slurry, measurement of immune activation (Interleukin-2) four hours after intake
  Interventions: Dietary Supplement: Barley hydrolyzed gluten 50 mg
- Placebo slurry (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo slurry

INTERVENTIONS:
Dietary Supplement: Wheat gluten 1000 mg — Nothing to add here
  Arms: Wheat gluten
Dietary Supplement: Barley gluten 1000 mg — Nothing to add here
  Arms: Barley gluten
Dietary Supplement: Barley gluten 50 mg — Nothing to add here
  Arms: Low dose barley gluten
Dietary Supplement: Barley hydrolyzed gluten 50 mg — Nothing to add here
  Arms: Low dose hydrolyzed barley gluten
Dietary Supplement: Placebo slurry — In slurry, measurement of immune activation (Interleukin-2) four hours after intake
  Arms: Placebo slurry

SUMMARY:
The study will compare the immune response in CeD patients to wheat and barley gluten at high doses (1 gram), and also investigate the reponses to low dose barley gluten and also hydrolyzed, malted barley and placebo. This will be done by five one-day challenges with intervals around four weeks.

DETAILED DESCRIPTION:
Celiac disease (CeD) is a common food-induced inflammatory disease of the small intestine caused by the ingestion of gluten from wheat, barley and rye. It is one of the most prevalent food hypersensitivities worldwide and affects 0.5-2.5% of the European population. The only effective treatment available is a strict lifelong gluten-free (GF) diet. GF products for CeD patients must not exceed the regulatory threshold of 20 mg/kg of gluten. Compliance of foods containing fermented or partially hydrolysed gluten is routinely assessed using the R5 competitive enzyme-linked immunosorbent assay (ELISA). However, this test does not adequately represent gluten immunogenicity in CeD patients. The overall objective of our ImmunoSafe-CeD proposal is to determine the CeD immunogenic activity of intact and partially hydrolysed gluten from wheat, rye and barley and develop improved comprehensive functional and analytical assays, including novel ELISAs and quantitative proteomics methods to ensure food safety for CeD patients. Thus, our objective is designed to directly address the needs of the CeD community about being reassured that GF products that contain partially hydrolysed gluten are safe and suitable for inclusion in their GF diet. By combining discovery proteomics and quantitative LC-MS/MS methods, improved reference materials for partially hydrolysed gluten, CeD-patient derived monoclonal antibodies and functional gluten-specific T-cell assays, we will provide a comprehensive and unique toolbox of novel and validated methods to detect gluten (both intact and partially hydrolysed) in foods for CeD patients.

This toolbox will close the current discrepancy between food analytical methods and CeD immunogenicity for the first time, because all methods will be matched to clinical pathophysiology assessed by food challenge in CeD patients. Our multidisciplinary consortium is built on previous highly successful collaborations and we are well-positioned to create even more synergies between us by exchanging materials, know-how and data. We expect to 1) better understand the role that the different glutens play in CeD pathogenesis, 2) develop easy-to-perform and reliable analytical tools (ELISA) that quantitate and predict immunogenicity (toxicity) of wheat, rye and barley products for CeD patients, and 3) define foods that CeD patients can tolerate despite being partly based on these processed grains

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30 kg/m2
* Biopsy verified celiac disease
* Pos gene test for HLA-DQ2.5 or DQ8
* Strict glutenfree diet for at least 24 months
* Clinical remission
* Sensitive to gluten by accidental intake
* Effective contraception if female in fertile age

Exclusion Criteria:

* Positive serology at screening
* Pregnant or lactating
* Other disease like Type 1 diabetes, cardiovascular disease, cancer, inflammatory bowel disease, thyroid or kidney disease
* On immunosuppressive drugs
* Smoking
* Food allergy including wheat allergy
* Acute infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Interleukin-2 in serum | 4 hours after intake
  Cytokine measurement by MSD Mesoscale

SECONDARY OUTCOMES:
GIP in urine 4 hours after challenge and feces 2 days after challenge | Four hours after challenge (urine) and 2 days after challenge (feces)
  Detection of gluten by test kits for BioMedal

CONTACTS AND LOCATIONS:
Overall Officials: Knut E A Lundin, PPhD, MD, Principal Investigator — Oslo University Hospital
Locations (2):
- Clinical Center for Celiac Disease and Autoimmunity, Mainz, Germany, Germany
- Dept of Gastroenterology, Oslo, Oslo County, Norway